CLINICAL TRIAL: NCT01868490
Title: Phase 1 Study of The Adoptive Immunotherapy for Solid Tumors Using Modified Autologous Cytokine-induced Killer Cells.
Brief Title: The Adoptive Immunotherapy for Solid Tumors Using Modified Autologous CIK Cells
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Principal Investigator, Adisak Wongkajornsilp, Pharmacology department, Faculty of medicine, Siriraj Hospital, Siriraj Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 215-3-2552; NCT01573455 (obsolete NCT alias)
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Cholangiocarcinoma; Neuroblastoma
Keywords: Cholangiocarcinoma; Cytokine induced killer cells; CIK; Treg; Th17; neuroblastoma
MeSH Terms: conditions — Cholangiocarcinoma; Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- drug (Experimental): single-group studies
  Interventions: Drug: cytokine induced killer cells

INTERVENTIONS:
Drug: cytokine induced killer cells — at least 10*9 CIK cells, IV on day 0, 14, 28

SUMMARY:
Cytokine-induced killer (CIK) cells exhibit high proliferation rate and cytotoxic activity in vitro. The major effector cells are the CD3+CD56+ subset. The cytolytic activity of CIK cells being independent of MHC restriction implies feasibility in using CIK cells allogeneic to the tumors. Experiments to block the MHC class-I and -II pathways on tumors-RNA transfected DCs showed that only MHC class-I blocking led to a significant reduction of heterogeneous CIK cells cytotoxicity after the co-culture. The safety of CIK cells was demonstrated by the lack of cytotoxicity toward autologous as well as allogeneic normal cells. Co-culture of CIK cells with dendritic cells (DCs) has been reported by us and others in a myriad of cancer (e.g., cholangiocarcinoma, osteosarcoma, glioblastoma multiforme, multiple myeloma, hepatocellular carcinoma, pancreatic carcinoma, renal & colon carcinoma, murine leukemia & lymphoma showing enhancement of anti-tumor cytotoxicity of CIK cell in all. The co-culture of CIK cells with DCs were reported to decrease the number of professional regulatory/ suppressor T cells (Treg, CD4+CD25+ cells) and decrease the secretion of IL-10, an immune suppressor cytokine, whereas the cytotoxic activity against target cells increased.

We have recently brought CIK cells through the preclinical phase (animal study) of human cholangiocarcinoma treatment. Cholangiocarcinoma (CCA), is a bile duct epithelial cancer endemic in the Northeast of Thailand, with an increasing incidence discernible in Europe and North America. Conventional treatments including surgery, chemotherapy, and radiation do not bring satisfactory survival due to anatomic location, presence of metastases, and high recurrent rates. These unsatisfactory outcomes urge to search innovative treatments such as immunotherapy. We reported the safety and efficacy of CIK cells in SCID mice model for cholangiocarcinoma. Several conditions of human CIK cells were examined using ex vivo cytotoxic assay and SCID mice pre-inoculated with human cholangiocarcinoma cells. We monitored the ex vivo cytotoxicity, tumor sizes and immunohistochemistry. Optimal tumor suppression was observed when CIK cells were pre-exposed to dendritic cells (DCs). Tumor-infiltrating human CD3+ cells were observed from day 2 - 14, but not in normal tissues elsewhere. These altogether indicated the specific homing of CIK cells to tumor mass. All animals did not exhibit any noticeable adverse reaction from the CIK treatments. The CD3+CD56+ cells are logical candidates for clinical trial while the DC-co-cultured CIK cells produced similar efficacy and more feasible for clinical application.

With a complete array of in vitro and in vivo study, the next rational step is moving forward to phase I/II clinical trials for a number of specified solid tumors (i.e., cholangiocarcinoma, osteosarcoma, and glioblastoma multiforme, nueroblastoma) using the optimized autologous CIK cells. Subjects without prior exposure to or weaned for at least 3 months from chemotherapy can be recruited to maintain the integrity of their immunological system, a critical factor for a successful immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 8 year-old, or allowance from their parent if younger than that.
2. Patient must have histologically or cytologically confirmed advanced cholangiocarcinoma or neuroblastoma by oncologist
3. The cancers have been failing to current treatment.
4. Patient is healthy by getting an Eastern Co-operative Oncology Group (ECOG) performances status of 0, 1 or 2.
5. Any of the following lab data

   a. Hematology:
   * Hb > 8 g/dl
   * Absolute neutrophil count (ANC) > 1,500 cells/mm3
   * Absolute lymphocyte count > 1,000 cells/mm3
   * Platelet > 100x109/L
6. Patient must have a life expectancy of at least 12 weeks by

   a. Biochemistry:
   * Serum total bilirubin < 3 mg/dl
   * Serum creatinine < 2 mg/dl
7. Patients will comply and provide written informed consent prior to enrollment into the study.

Exclusion Criteria:

1. Patients received chemotherapy within 4 weeks before study entry.
2. Active uncontrolled infection
3. Concurrent anti-cancer treatment in another investigational trial, including immunotherapy in last 30 days
4. Pregnant or lactating woman, or women of child bearing potential or less than one year after menopause (unless surgically sterile) with urine pregnancy test positive
5. Concurrent steroid therapy

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-04-17 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
MRI scan for monitoring of tumor size and CIK cell-homing, Fluorescence-activated cell sorting (FACS) analysis | 6 weeks

SECONDARY OUTCOMES:
Survival rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Adisak Wongkajornsilp, M.D., Ph.D., Principal Investigator — Mahidol University
Locations (2):
- Thailand (2):
  - Siriraj Clinical Research Center, Siriraj Hospital, Bangkoknoi, Bangkok
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok

IPD SHARING:
Plan to Share IPD: No